CLINICAL TRIAL: NCT00476723
Title: Generation of HBV-specific T-cell Immunity in Individuals With HIV/HBV Co-infection Receiving HBV-active Antiretroviral Therapy
Brief Title: HBV-specific T-cell Immunity in Individuals With HIV/HBV Co-infection
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Kirby Institute (Other Government); Ministry of Health, Thailand (Other Government)
Responsible Party: Prof. Kiat Ruxrungtham, HIV-NAT
Other Study IDs: HIV-NAT 032
Record Dates: First submitted 2006-11-15; First posted 2007-05-22 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: HIV; Hepatitis-B
Keywords: HIV infection; Hepatitis coinfection
MeSH Terms: conditions — Hepatitis B; HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: HIV/Hepatitis coinfected patients who use at least one hepatitis activity drug or medications

SUMMARY:
The trial will randomise HIV/HBV co-infected individuals to different HBV-active antiretroviral therapy treatment regimens.

DETAILED DESCRIPTION:
Longitudinal study of circulating and intra-hepatic HBV-specific T-cell immunity in the setting of a randomised, controlled, international, multi-centre outpatient trial. The trial will randomise HIV/HBV co-infected individuals to different HBV-active antiretroviral therapy treatment regimens.

Study population: Patients with HIV/HBV co-infection who are naive to HIV/HBV therapy, have detectable HBV viremia and are willing to start antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* hepatitis-B co-infected
* HBV/HIV therapy naive
* >18 years of age

Exclusion Criteria:

Unable to sign consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV/Hepatitis B coinfected patients using at least one hepatitis active medications in HAART regimen
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To characterize circulating and intra-hepatic anti-HBV T-cell responses longitudinally in HIV-1/HBV co-infected individuals, following effective anti-HBV therapy | 48 weeks

SECONDARY OUTCOMES:
To identify novel CD4 and CD8 T cell HBV epitopes associated with HBV clearance. | 48 weeks
To identify emergence of cytotoxic T lymphocyte (CTL) "escape" mutants following anti-HBV therapy | 48 weeks
To determine the effect of HIV-1 co-infection and anti-HBV T-cell responses on clearance of free virions and HBV reservoirs using viral dynamic parameters and direct quantification of HBV hepatic reservoirs | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, MSc, Principal Investigator — HIV-NAT, The Thai Red Cross AIDS Research Centre
Locations (1):
- HIV-NAT, Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org